CLINICAL TRIAL: NCT06173648
Title: Histopathological Evaluation of the Periodontal Ligament and Cementum of Extracted Teeth Subjected to Laser Ablation With Indocyanine Green.
Brief Title: Histopathological Evaluation of the Periodontal Ligament Subjected to Laser Ablation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAO Group, Inc. (Industry)
Collaborators: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70009423.2.0000.5539
Record Dates: First submitted 2023-11-16; First posted 2023-12-18 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Single study group requiring extraction of mandibular incisors for other reasons. Controls selected from among the extraction candidates were not subject to exposure to the laser and ICG solution, but to all other aspects of the pulpectomy procedure. Remaining teeth had the laser and ICG exposure added to the treatment regimen. Treated and control specimens then extracted, prepared, stained, and examined for histological morphological condition of the periodontal ligament, cementum, and collagen attached to the external surface of the extracted tooth root.
Masking Description: Blinding occurred when analyzing the histological and morphological results. Blinded assessor provided a rating of the samples on an individual basis, not knowing if the sample was from a treated or control tooth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- All Study Participants. (Experimental): Single study group that requires extraction of mandibular incisors for other reasons. Teeth are accessed, subject to filing, pulp extirpation, and treated with endodontic solutions. Some teeth of the participants are then subject to study intervention consisting of an ICG solution into the root followed by laser exposure of the solution in situ. After laser exposure, the pulp chamber and roots are rinsed then mechanically extracted. Other teeth of some participants will not be subject to the ICG and laser intervention, but will proceed to the final rinse and extraction. After extraction, specimens are fixed, stained, and mounted for visual examination under a microscope. Images of tissue are captured for documentation. Samples are examined for histological and morphological condition of the periodontal ligament, cementum, and collagen attached to the external surface of the extracted tooth root.
  Interventions: Device: Laser and ICG solution.

INTERVENTIONS:
Device: Laser and ICG solution. — Intervention consists of addition of a combined laser absorption solution and infrared diode laser. The solution is introduced into the prepared pulp chamber and root canals, allowed to dwell for 1 minute, followed by exposure to the laser energy delivered via a fiber optic introduced into the root canal, and while activating the laser at 2.5 watts of optical output with a pulse duration of 100 msec and a pulse gap of 300 msec, the solution and residual structures in the root and pulp chamber are exposure over the course of 30 seconds, moving and relocating the fiber tip throughout the canals and chamber during that time. The laser is halted and a wait time of 30 seconds is applied. The laser fiber is then reintroduced and another 30 second exposure, repeating the same settings and technique.
  Other Names: Leonardo Diode Laser and LEAP Laser Absorption Solution

SUMMARY:
Laser Ablation therapy (LA) using an 810nm diode laser and Indocyanine Green (ICG) solution, which efficiently absorbs laser energy and increases the effectiveness of tissue removal. Intracanal heating can potentially cause damage to structures outside the tooth root. The study was to observe possible changes in the periodontal ligament and cementum resulting outside the root using this treatment. Histological and morphological examination of extracted cementum, ligament, and collagen post-exposure showed no difference in these structures vs. non-treated controls.

DETAILED DESCRIPTION:
Laser Ablation therapy (LA) using 810nm diode laser and Indocyanine Green (ICG) solution which efficiently absorbs laser energy and the increased temperature results in an instantaneous flame that chars tissue and microbes. Intracanal heating can potentially cause damage to cementum structure and periodontal tissues. The objective of this study is to observe possible changes in the periodontal ligament and cementum resulting from the use of LA with ICG as an adjuvant therapy to endodontic treatment. Ten patients with lower incisors requiring extraction will be selected. Before extraction, chemical-mechanical root canal preparation will be carried out with a single file reciprocating system (35/04) and 2.5% sodium hypochlorite solution. Then, the canals will be dried and filled with 0.05% ICG, which will remain in place for 1 minute (pre-irradiation time). For the test group, a #20 laser fiber will be inserted into the root canal to the working length. The 810 nm wavelength infrared diode laser is activated with a power of 2.5W, an interval of 300 ms, and a duration of 100 ms. After activation commences, circular movements are made for a period of 30 seconds together with the fiber removal movement. After the first activation, there is a 30-second pause and a new 30-second activation cycle will then be performed in the same way as the previous one. After treatment, the tooth element will be extracted and the apical third of the root with the periodontal ligament is processed for histological analysis using hematoxylin-eosin and picrosirius red staining to evaluate the morphological structures. Two teeth extracted without treatment will be used as controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Requiring at a least one mandibular incisor to be extracted.

Exclusion Criteria:

* Evidence of periodontal disease anywhere in the mouth beyond the apical third of any tooth.
* Mandibular canines that do not require extraction.
* Presence of other dental or oral conditions of any type that require immediate intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unicesumar Clinic, Maringá, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no issues with participant wash-out after initial acceptance into the study.
Units Other Than Participants: Mandibular Incisor Teeth
Groups:
- Teeth Exposed to Laser and ICG Solution.: Single study group that requires extraction of mandibular incisors for other reasons. Teeth will be accessed, subject to mechanical file, pulp extirpation, and treated with endodontic solutions. Teeth will then be exposed to the ICG solution followed by laser exposure of the ICG solution in situ. After laser exposure, the pulp chamber and roots will be rinsed and then the tooth mechanically extracted. After extraction, tissue specimens will be prepared of the root portion of the extracted tooth, fixed, stained, and mounted for visual examination under a microscope. Images of the microscopic images will be captured for documentation. The samples will be examined for the histological and morphological condition of the periodontal ligament, cementum, and collagen attached to the external surface of the extracted tooth root. These tissue types were graded based on the extent of damage or destruction observed.
  Laser and ICG solution.: Intervention consists of addition of laser absorption solution and infrared diode laser. The solution is introduced into pulp chamber and root canals, dwells for 1 minute, followed by exposure to the laser delivered via optical fiber introduced into the root canal, activating the laser at 2.5W optical output, pulse duration of 100msec and pulse gap of 300msec, with laser emissions totaling 30s, moving and relocating the fiber during the exposure. The laser is halted, a 30s wait, then solution and laser is repeated.
Period: Overall Study
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Started | 10; 12 Mandibular Incisor Teeth (2 units were not subject to the interventional aspect, but were utilized as control teeth.)
Completed | 10; 12 Mandibular Incisor Teeth (2 units were not subject to the interventional aspect, but were utilized as control teeth.)
Not Completed | 0; 0 Mandibular Incisor Teeth

BASELINE CHARACTERISTICS:
Population: A total of 10 participants were involved in the study. All 10 participants contributed 1 tooth to the interventional group. Additionally, 2 of the participants contributed an additional tooth that was subject to the control treatment conditions.
Units Other Than Participants: Teeth
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Number analyzed (Participants) | 10
Number analyzed (Teeth) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 10

OUTCOME MEASURES:

1. Primary Outcome: Cell Count of Inflammatory Infiltrate Per Cross-Sectional Area at 400X Magnification
Description: Count the number of inflammatory cells within a cross-sectional area viewed under 400X magnification, comparing the difference in the quantity of inflamed cells reacting to injury to the tissues resulting from the investigational treatment, as compared a count of inflamed cells reacting to the control treatment.
Time Frame: 28 days after intervention.
Population: Mandibular incisor teeth
Measure: Mean (Standard Deviation); unit: Cells / 0.1 mm^2
Units Other Than Participants: Teeth
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Number analyzed (Participants) | 10
Number analyzed (Teeth) | 12
Cells / 0.1 mm^2
  Intervention: number analyzed (Teeth) | 10
  Intervention | 10.3 (1.79)
  Control: number analyzed (Participants) | 2
  Control: number analyzed (Teeth) | 2
  Control | 10.5 (0.2)

2. Primary Outcome: Gap Distance of Inflammatory Resorption Between Inflamed Tissue and Root Surface
Description: Measurement of the gap between the edge of the inflamed tissue and the root surface, measured in microns using computer software to measure the gap of magnified tissue samples, comparing samples from teeth treated with the intervention compared to teeth receiving the control treatment.
Time Frame: 28 days after intervention.
Population: Mandibular incisor teeth
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: Teeth
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Number analyzed (Participants) | 10
Number analyzed (Teeth) | 12
micrometer
  Intervention: number analyzed (Teeth) | 10
  Intervention | 0 (0)
  Control: number analyzed (Participants) | 2
  Control: number analyzed (Teeth) | 2
  Control | 0 (0)

3. Primary Outcome: Mean Ligament Thickness of the Periodontal Ligament
Description: Measurement of the thickness of the periodontal ligament, measured in microns using computer software to measure the thickness of periodontal ligament within the magnified tissue samples, comparing samples from teeth treated with the intervention compared to teeth receiving the control treatment.
Time Frame: 28 days after intervention.
Population: Mandibular incisor teeth
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: Teeth
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Number analyzed (Participants) | 10
Number analyzed (Teeth) | 12
micrometer
  Intervention: number analyzed (Teeth) | 10
  Intervention | 173.55 (14.33)
  Control: number analyzed (Participants) | 2
  Control: number analyzed (Teeth) | 2
  Control | 178.8 (6.66)

4. Secondary Outcome: Gap Distance of Inflammatory Resorption Between Cementum and Alveolar Bone
Description: Measurement of the gap between the edge of the tooth cementum and the adjacent alveolar bone, measured in microns using computer software to measure the gap of magnified tissue samples, comparing samples from teeth treated with the intervention compared to teeth receiving the control treatment.
Time Frame: 28 days after intervention.
Population: Mandibular incisor teeth
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: Teeth
Arm/Group | Teeth Exposed to Laser and ICG Solution.
Number analyzed (Participants) | 10
Number analyzed (Teeth) | 12
micrometer
  Intervention: number analyzed (Teeth) | 10
  Intervention | 0 (0)
  Control: number analyzed (Participants) | 2
  Control: number analyzed (Teeth) | 2
  Control | 0 (0)

ADVERSE EVENTS:
Time Frame: 14 days post-treatment
Description: Adverse event was evaluated on the day of treatment, and at a 14-day post treatment follow-up.
Groups:
- Control Teeth Not Exposed to Laser and ICG Solution.: Single study group that requires extraction of mandibular incisors for other reasons. Teeth will be accessed, subject to mechanical file, pulp extirpation, and treated with endodontic solutions. The pulp chamber and roots will be rinsed and then the tooth mechanically extracted. After extraction, tissue specimens will be prepared of the root portion of the extracted tooth, fixed, stained, and mounted for visual examination under a microscope. Images of the microscopic images will be captured for documentation. The samples will be examined for the histological and morphological condition of the periodontal ligament, cementum, and collagen attached to the external surface of the extracted tooth root. These tissue types were graded based on the extent of damage or destruction observed.
Arm/Group | Teeth Exposed to Laser and ICG Solution. | Control Teeth Not Exposed to Laser and ICG Solution.
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 0/10 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT06173648/Prot_SAP_000.pdf